CLINICAL TRIAL: NCT03537638
Title: Effectiveness and Cost-effectiveness of a Multicomponent Strategy to Implement a Clinical Practice Guideline and Improve Health Outcomes in People With Systemic Lupus Erythematosus
Brief Title: Multicomponent Strategy to Implement a Clinical Practice Guideline and Improve Health Outcomes in People With SLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Servicio Canario de Salud (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: PI15/01377
Record Dates: First submitted 2018-04-16; First posted 2018-05-25 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2020-10

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Lupus; Quality of life; Multicomponent intervention; Clinical Practice Guideline; Computerized clinical decision support system; Activity
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multicomponent Intervention (Experimental): Rheumatologist and internist receive a multicomponent intervention
  Interventions: Behavioral: Multicomponent intervention
- Control (No Intervention): Rheumatologist and internist provide the usual care

INTERVENTIONS:
Behavioral: Multicomponent intervention — Intervention to rheumatologist and internist responsible for the care of patients with SLE. Implementation multicomponent intervention consisting of: educational component, a computerized clinical decision support system developed from the clinical practice guide - SLE and automated feedback integrated into the electronic medical record system.
  Arms: Multicomponent Intervention

SUMMARY:
Principal objective: To produce scientific knowledge on the effectiveness and cost-effectiveness of a multicomponent intervention for knowledge transfer and implementing a Clinical Practice Guideline (CPG) for Systemic Lupus Erythematosus (SLE), formed by an educative intervention, an computerized clinical decision support system (SADC), complemented by an automated feedback built into the electronic clinical record.

Secondary objectives will be previously developed: 1) the analysis of medical practice variations along the care of SLE patients in the Canary Islands Health Service (SCS); 2) the best available scientific evidence to support the optimal development of the SADC; 3) the context and the barriers to innovation implementation in the SCS; and 4) the development of the contents for the implementation strategy, including the SADC and the automated feedback.

Methods for the main objective: The main objective will be assessed under an open, multicentric and randomized (by clusters) clinical trial, in the SCS. The multicomponent intervention will be compared to the usual procedures for CPG dissemination. The main measure will be the self-perceived activity of SLE rated by the SLAQ scale. Self-perceived health related quality of life (HRQoL) data will be obtained by means of the questionnaire EQ-5D-5L , to estimate a cost-effectiveness ratio.

Methods for secondary objectives: The rest of the objectives will be developed by a mix of quantitative and qualitative research methods to allow adapting the design, development and execution of the intervention to the characteristics of the context.

ELIGIBILITY:
Inclusion Criteria:

* Patients:

Adults (older than 18 years) diagnosed with SLE of any seriousness and situation (active, remission or clinically quiescent and serologically active), who agree to participate and sign informed consent.

* Health professionals:

Physicians specialized in rheumatology or internal medicine that include in their quotas a minimum of 30 patients with eligible SLE.

Exclusion Criteria:

* Patients:

SLE limited to the skin, advanced chronic kidney disease (dialysis or renal transplant); Mental illnesses and / or sensory or cognitive deficits; or participating in extension or follow-up studies of another RCT (possible change in follow-up guidelines). Participants in observational studies may be included as they do not change usual practice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2020-10-19 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change of self-perceived activity of the SLE | 18 months
  Disease activity self-reported by the patient using the Systemic Lupus Erythematosus Activity (SLAQ) Questionnaire

SECONDARY OUTCOMES:
Change in professional's knowledge about SLE management | 18 months
  Acquired knowledges assessed by a questionnaire designed ad hoc
Change in self-perceived health-related quality of life | 18 months
  Self-perceived health-related quality of life using EQ-5D - 5L questionnaire
Change in self-perceived health-related quality of life | 18 months
  Self-perceived health-related quality of life using LupusQol questionnaire
Patient's perception of their participation in decision making | 18 months
  Patient's perception of clinician facilitation and decision-making process using the Shared Decision-Making (SDM-Q-9) Questionnaire
Professional's attitude to partnership with the patient for shared decision making | 18 months
  Professionals' attitudes towards shared decision making assessed by the Leeds Attitude Towards Concordance II Scale (LATCon II)
Professionals' adherence to CPG-SLE recommendations | 18 months
  Degree of professional adherence to recommendations will be determined through data collection from clinical records in terms of percentage of patients with adequate treatment according to SLE-CPG recommendations

CONTACTS AND LOCATIONS:
Overall Officials: María de Mar Trujillo Martin, PhD, Principal Investigator — Servicio de Evaluación del Servicio Canario de la Salud
Locations (1):
- Servicio de Evaluación del Servicio Canario de la Salud, Santa Cruz de Tenerife, Spain

REFERENCES:
- [Background] Serrano-Aguilar P, Kovacs FM, Cabrera-Hernandez JM, Ramos-Goni JM, Garcia-Perez L. Avoidable costs of physical treatments for chronic back, neck and shoulder pain within the Spanish National Health Service: a cross-sectional study. BMC Musculoskelet Disord. 2011 Dec 21;12:287. doi: 10.1186/1471-2474-12-287. PMID 22188790
- [Background] Ostbye T, Yarnall KS, Krause KM, Pollak KI, Gradison M, Michener JL. Is there time for management of patients with chronic diseases in primary care? Ann Fam Med. 2005 May-Jun;3(3):209-14. doi: 10.1370/afm.310. PMID 15928223
- [Background] Zhu TY, Tam LS, Li EK. Cost-of-illness studies in systemic lupus erythematosus: A systematic review. Arthritis Care Res (Hoboken). 2011 May;63(5):751-60. doi: 10.1002/acr.20410. PMID 21557530
- [Background] Lerang K, Gilboe IM, Gran JT. Differences between rheumatologists and other internists regarding diagnosis and treatment of systemic lupus erythematosus. Rheumatology (Oxford). 2012 Apr;51(4):663-9. doi: 10.1093/rheumatology/ker318. Epub 2011 Dec 7. PMID 22157467
- [Background] Bertsias G, Ioannidis JP, Boletis J, Bombardieri S, Cervera R, Dostal C, Font J, Gilboe IM, Houssiau F, Huizinga T, Isenberg D, Kallenberg CG, Khamashta M, Piette JC, Schneider M, Smolen J, Sturfelt G, Tincani A, van Vollenhoven R, Gordon C, Boumpas DT; Task Force of the EULAR Standing Committee for International Clinical Studies Including Therapeutics. EULAR recommendations for the management of systemic lupus erythematosus. Report of a Task Force of the EULAR Standing Committee for International Clinical Studies Including Therapeutics. Ann Rheum Dis. 2008 Feb;67(2):195-205. doi: 10.1136/ard.2007.070367. Epub 2007 May 15. PMID 17504841
- [Background] Sidorenkov G, Haaijer-Ruskamp FM, de Zeeuw D, Denig P. A longitudinal study examining adherence to guidelines in diabetes care according to different definitions of adequacy and timeliness. PLoS One. 2011;6(9):e24278. doi: 10.1371/journal.pone.0024278. Epub 2011 Sep 8. PMID 21931669
- [Background] Perez X, Wisnivesky JP, Lurslurchachai L, Kleinman LC, Kronish IM. Barriers to adherence to COPD guidelines among primary care providers. Respir Med. 2012 Mar;106(3):374-81. doi: 10.1016/j.rmed.2011.09.010. Epub 2011 Oct 13. PMID 22000501
- [Background] Kastner M, Bhattacharyya O, Hayden L, Makarski J, Estey E, Durocher L, Chatterjee A, Perrier L, Graham ID, Straus SE, Zwarenstein M, Brouwers M. Guideline uptake is influenced by six implementability domains for creating and communicating guidelines: a realist review. J Clin Epidemiol. 2015 May;68(5):498-509. doi: 10.1016/j.jclinepi.2014.12.013. Epub 2015 Jan 10. PMID 25684154
- [Background] Cabana MD, Rand CS, Powe NR, Wu AW, Wilson MH, Abboud PA, Rubin HR. Why don't physicians follow clinical practice guidelines? A framework for improvement. JAMA. 1999 Oct 20;282(15):1458-65. doi: 10.1001/jama.282.15.1458. PMID 10535437
- [Background] Jacobs SR, Weiner BJ, Bunger AC. Context matters: measuring implementation climate among individuals and groups. Implement Sci. 2014 Apr 17;9:46. doi: 10.1186/1748-5908-9-46. PMID 24742308
- [Background] Francke AL, Smit MC, de Veer AJ, Mistiaen P. Factors influencing the implementation of clinical guidelines for health care professionals: a systematic meta-review. BMC Med Inform Decis Mak. 2008 Sep 12;8:38. doi: 10.1186/1472-6947-8-38. PMID 18789150
- [Background] Grimshaw JM, Eccles MP, Lavis JN, Hill SJ, Squires JE. Knowledge translation of research findings. Implement Sci. 2012 May 31;7:50. doi: 10.1186/1748-5908-7-50. PMID 22651257
- [Background] Sketris IS, Langille Ingram EM, Lummis HL. Strategic opportunities for effective optimal prescribing and medication management. Can J Clin Pharmacol. 2009 Winter;16(1):e103-25. Epub 2009 Jan 30. PMID 19182305
- [Background] Giguere A, Legare F, Grimshaw J, Turcotte S, Fiander M, Grudniewicz A, Makosso-Kallyth S, Wolf FM, Farmer AP, Gagnon MP. Printed educational materials: effects on professional practice and healthcare outcomes. Cochrane Database Syst Rev. 2012 Oct 17;10(10):CD004398. doi: 10.1002/14651858.CD004398.pub3. PMID 23076904
- [Background] Shojania KG, Jennings A, Mayhew A, Ramsay CR, Eccles MP, Grimshaw J. The effects of on-screen, point of care computer reminders on processes and outcomes of care. Cochrane Database Syst Rev. 2009 Jul 8;2009(3):CD001096. doi: 10.1002/14651858.CD001096.pub2. PMID 19588323
- [Background] Baker R, Camosso-Stefinovic J, Gillies C, Shaw EJ, Cheater F, Flottorp S, Robertson N. Tailored interventions to overcome identified barriers to change: effects on professional practice and health care outcomes. Cochrane Database Syst Rev. 2010 Mar 17;(3):CD005470. doi: 10.1002/14651858.CD005470.pub2. PMID 20238340
- [Background] Gillaizeau F, Chan E, Trinquart L, Colombet I, Walton RT, Rege-Walther M, Burnand B, Durieux P. Computerized advice on drug dosage to improve prescribing practice. Cochrane Database Syst Rev. 2013 Nov 12;2013(11):CD002894. doi: 10.1002/14651858.CD002894.pub3. PMID 24218045
- [Background] Murphy EV. Clinical decision support: effectiveness in improving quality processes and clinical outcomes and factors that may influence success. Yale J Biol Med. 2014 Jun 6;87(2):187-97. eCollection 2014 Jun. PMID 24910564
- [Background] Ramallo-Farina Y, Garcia-Perez L, Castilla-Rodriguez I, Perestelo-Perez L, Wagner AM, de Pablos-Velasco P, Dominguez AC, Cortes MB, Vallejo-Torres L, Ramirez ME, Martin PP, Garcia-Puente I, Salinero-Fort MA, Serrano-Aguilar PG; INDICA team. Effectiveness and cost-effectiveness of knowledge transfer and behavior modification interventions in type 2 diabetes mellitus patients--the INDICA study: a cluster randomized controlled trial. Implement Sci. 2015 Apr 9;10:47. doi: 10.1186/s13012-015-0233-1. PMID 25880498
- [Background] Roshanov PS, Fernandes N, Wilczynski JM, Hemens BJ, You JJ, Handler SM, Nieuwlaat R, Souza NM, Beyene J, Van Spall HG, Garg AX, Haynes RB. Features of effective computerised clinical decision support systems: meta-regression of 162 randomised trials. BMJ. 2013 Feb 14;346:f657. doi: 10.1136/bmj.f657. PMID 23412440
- [Background] Lobach D, Sanders GD, Bright TJ, Wong A, Dhurjati R, Bristow E, Bastian L, Coeytaux R, Samsa G, Hasselblad V, Williams JW, Wing L, Musty M, Kendrick AS. Enabling health care decisionmaking through clinical decision support and knowledge management. Evid Rep Technol Assess (Full Rep). 2012 Apr;(203):1-784. PMID 23126650
- [Background] Hoffmann TC, Montori VM, Del Mar C. The connection between evidence-based medicine and shared decision making. JAMA. 2014 Oct 1;312(13):1295-6. doi: 10.1001/jama.2014.10186. No abstract available. PMID 25268434
- [Background] Elwyn G, Frosch D, Thomson R, Joseph-Williams N, Lloyd A, Kinnersley P, Cording E, Tomson D, Dodd C, Rollnick S, Edwards A, Barry M. Shared decision making: a model for clinical practice. J Gen Intern Med. 2012 Oct;27(10):1361-7. doi: 10.1007/s11606-012-2077-6. Epub 2012 May 23. PMID 22618581
- [Background] Serrano-Aguilar P, Trujillo-Martin Mdel M, Perez de la Rosa A, Cuellar-Pompa L, Saavedra-Medina H, Linertova R, Perestelo-Perez L, Perez-Ramos J, Rivero-Santana A; Spanish SLE CPG Development Group. Patient participation in a Clinical Guideline Development for Systemic Lupus Erythematosus. Patient Educ Couns. 2015 Sep;98(9):1156-63. doi: 10.1016/j.pec.2015.05.022. Epub 2015 Jun 11. PMID 26095343
- [Background] Politi MC, Wolin KY, Legare F. Implementing clinical practice guidelines about health promotion and disease prevention through shared decision making. J Gen Intern Med. 2013 Jun;28(6):838-44. doi: 10.1007/s11606-012-2321-0. Epub 2013 Jan 10. PMID 23307397
- [Background] Loya SR, Kawamoto K, Chatwin C, Huser V. Service oriented architecture for clinical decision support: a systematic review and future directions. J Med Syst. 2014 Dec;38(12):140. doi: 10.1007/s10916-014-0140-z. Epub 2014 Oct 18. PMID 25325996
- [Background] Panzarasa S, et al.Technical Solutions for Integrating Clinical Practice Guidelines with Electronic Patient Records. Volume 5943 of LNAI. Springer-Verlag 2010;141 -154
- [Background] Kawamoto K, Del Fiol G, Orton C, Lobach DF. System-agnostic clinical decision support services: benefits and challenges for scalable decision support. Open Med Inform J. 2010;4:245-54. doi: 10.2174/1874431101004010245. Epub 2010 Dec 14. PMID 21603281
- [Derived] Trujillo-Martin MM, Ramallo-Farina Y, Del Pino-Sedeno T, Rua-Figueroa I, Trujillo-Martin E, Vallejo-Torres L, Imaz-Iglesia I, Sanchez-de-Madariaga R, de Pascual-Medina AM, Serrano-Aguilar P; SLE-CPG-Implementation Group. Effectiveness and cost-effectiveness of a multicomponent intervention to implement a clinical practice guideline for systemic lupus erythematosus: protocol for a cluster-randomized controlled trial. BMC Health Serv Res. 2019 Nov 1;19(1):783. doi: 10.1186/s12913-019-4589-9. PMID 31675957